CLINICAL TRIAL: NCT01823146
Title: Oxytocin and Aging: Neuro-Behavioral Effects on Social Cognition and Prosocial Behavior
Brief Title: Oxytocin's Effect on Socioemotional Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 39-2013; UL1TR000064 (NIH)
Record Dates: First submitted 2013-03-25; First posted 2013-04-04 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2015-10

CONDITIONS: Aging
Keywords: oxytocin; socioemotional functioning; trust; amygdala; aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin spray (Experimental): single dose of 24 IU oxytocin, self-administered intranasally (IN)
  Interventions: Drug: Oxytocin spray
- Placebo spray (Placebo Comparator): single dose of 24 IU placebo (same solution as oxytocin spray but without oxytocin), self-administered intranasally (IN)
  Interventions: Drug: Placebo spray

INTERVENTIONS:
Drug: Oxytocin spray — single dose of 24 IU oxytocin, self-administered intranasally (IN)
  Arms: Oxytocin spray
Drug: Placebo spray — single dose of 24 IU placebo (same solution as oxytocin spray but without oxytocin), self-administered intranasally (IN)
  Arms: Placebo spray

SUMMARY:
This study will investigate the extent to which intranasal oxytocin affects changes in social decision making and evaluations of others. Oxytocin is a hormone that naturally occurs in the body and the brain and has been shown to be relevant for many behaviors, particularly in social situations. Research on the effects of oxytocin in aging is very scarce; therefore, the purpose of this research project is to determine the effects of oxytocin on socioemotional aging.

DETAILED DESCRIPTION:
In order to demonstrate oxytocin as a causal mechanism in socioemotional aging, the investigators propose to temporarily elevate oxytocin levels and then measure activity in the brain while participants engage in socially relevant tasks. Participants in this study will be randomly assigned (much like flipping a coin) to receive either a single administration of oxytocin or a placebo (a substance that looks like the oxytocin but does not have any active drug). Neither participants nor the investigator will know to which condition each participant is assigned. Prior to being enrolled into the study a screening to determine eligibility will be conducted. Once the screening visit is completed and it has been determined that subjects can be randomized into the study, an appointment will be scheduled for the full study visit.

The purpose of the screening is to determine whether the individual is eligible for participation in the study and will consist of a series of questions about demographics and health history, two saliva samples, two short tasks, blood test, and brief meeting with a licensed clinician to ensure that it is safe for the individual to take part in the magnetic resonance imaging (MRI) and drug administration.

The study visit will comprise two collections of saliva for laboratory tests prior to and following the oxytocin administration in order to measure levels of the hormone in the body at baseline and after the spray. Saliva samples will also allow for an examination of how oxytocin-related genes may impact cognition and behavior during study tasks. Participants will work on various social tasks while in the MRI scanner, and response accuracy, response time, and brain activity will be recorded. After the scan, participants will complete a series of brief questionnaires on paper and on the computer.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30 years or 63-85 years
* English fluency
* Caucasian
* Right-handed

Exclusion Criteria:

* Pregnant or possibly pregnant
* Breastfeeding
* Claustrophobia
* Currently on vasoconstrictors, pseudoephedrine or antidiuretic medication
* Large pieces of metal in the body, particularly in the face or neck
* Piercings or metal implants that cannot be removed from the body
* Surgery on the brain or any prior serious brain damage or disease
* Dementia or severe cognitive disorders
* History of hyponatremia, Syndrome of Inappropriate Antidiuretic Hormone, psychogenic polydipsia, or motion disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie C Ebner, PhD, Principal Investigator — University of Florida, Department of Psychology
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 08/2013 and 09/2014. Recruitment phone calls were conducted at the Social-Cognitive and Affective Development Lab at University of Florida.
Groups:
- Placebo Spray: single dose of 24 IU saline, self-administered intranasally (IN). This is an identical solution to the oxytocin spray but without the oxytocin.
Period: Overall Study
Arm/Group | Oxytocin Spray | Placebo Spray
Started | 55 | 51
Completed | 53 | 49
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Spray: single dose of 24 IU saline, self-administered intranasally (IN)
- Total: Total of all reporting groups
Arm/Group | Oxytocin Spray | Placebo Spray | Total
Number analyzed (Participants) | 55 | 51 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 26 | 60
  >=65 years | 21 | 25 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 27 | 24 | 51
Region of Enrollment [Number; unit: participants]
  United States | 55 | 51 | 106

OUTCOME MEASURES:

1. Primary Outcome: Extent of Trust Behavior
Description: Average amount of monetary units invested in the context of the Trust/Lottery Game.
  The theoretical range was 0 to 72 monetary units across all 24 trials. Participants invested in 12 social (human person) and 12 non-social (computer) trials.The mean average amount of monetary units invested was calculated for social and non-social trials separately.
Time Frame: 45 minutes after drug/placebo administration
Population: All study participants who had undergone the screening as well as the full visit (n = 102).
Measure: Mean (Standard Error); unit: monetary units
Arm/Group | Oxytocin Spray | Placebo Spray
Number analyzed (Participants) | 53 | 49
monetary units
  non-social trials | 39.03 (2.55) | 44.42 (2.54)
  social trials | 45.11 (1.86) | 46.06 (2.47)

2. Secondary Outcome: Meta-Mood
Description: Mean self-reported level of meta-mood for the two subscales attention to feelings and clarity of feelings. Response scale ranged from 1 to 5, with higher scores indicating more attention to feelings and greater clarity of feelings, respectively. The mean score for the subscales were calculated.
Time Frame: 2.5 hours after drug/placebo administration
Population: All study participants who had undergone the screening as well as the full visit (n = 102).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin Spray | Placebo Spray
Number analyzed (Participants) | 53 | 49
units on a scale
  n = 24 older men (63 to 85 years) | 3.38 (.18) | 2.977 (.19)
  n = 30 older women (63 to 85 years) | 3.23 (.18) | 3.63 (.17)
  n = 25 young men (18 to 30 years) | 3.54 (.17) | 3.58 (.20)
  n = 23 young women (18 to 30 years) | 4.04 (.19) | 3.68 (.21)

3. Secondary Outcome: Functional Connectivity (Resting fMRI)
Description: The functional connectivity (strength measure in units on a scale) between amygdala and medial prefrontal cortex was measured via a resting functional magnetic resonance imaging scan (participants looked at a fixation cross while images of their brain at rest were taken). Functional connectivity is the connectivity between brain regions (i.e., amygdala and medial prefrontal cortex) that share functional properties. It is defined as the temporal correlation between spatially remote neurophysiological events, expressed as deviation from statistical independence across these events in distributed neuronal groups and areas. A mean of this correlation (connectivity strength) was computed and transformed into z-scores (r to z transformation). The z-scores ranged from -2 to +2 with higher scores representing a greater resting-state functional connectivity.
Time Frame: 1.5 hours after oxytocin/placebo administration
Population: All study participants who had undergone the screening as well as the full visit and had reliable resting fMRI scan data (e.g., low extent of head motion) (n = 79).
Measure: Least Squares Mean (95% Confidence Interval); unit: z-scores
Arm/Group | Oxytocin Spray | Placebo Spray
Number analyzed (Participants) | 40 | 39
z-scores | 0.58 [0.49 to 0.66] | 0.48 [0.39 to 0.57]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo Spray: single dose of 24 IU saline, self-administered intranasally (IN)
  Placebo spray: single dose of 24 IU saline, self-administered intranasally (IN)
Arm/Group | Oxytocin Spray | Placebo Spray
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/51
Other Adverse Events (participants affected / at risk) | 0/55 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No